CLINICAL TRIAL: NCT06540560
Title: Exploring Patient Treatment Preferences for Chronic Pelvic Pain: A Mixed Methods Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sara Till, MD, MPH, Assistant Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00253781; 1K23HD099283-01A1 (NIH)
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pelvic Pain
Keywords: Structured interview; Questionnaires; Web-based educational program

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My Pelvic Plan (Experimental): This is a web-based self-guided program.
  Interventions: Behavioral: My Pelvic Plan website

INTERVENTIONS:
Behavioral: My Pelvic Plan website — Following the baseline interview, participants will receive a link to a web-based self-guided program and have access for two weeks "My Pelvic Plan" that combines education on several individual conditions that often contribute to CPP, and will include instruction on cognitive and behavioral restructuring, self-administration of acupressure, engaging in physical activity, and a brief introduction to pelvic floor physical therapy techniques. Subsequent to this, participants will then complete another brief questionnaire after a two-week interval. This questionnaire will focus on willingness to consider specific treatment modalities, credibility/expectancy for specific treatment modalities, and a brief measure assessing self-efficacy for managing symptoms.

SUMMARY:
This research is studying what things change the way people think about treatment for chronic pelvic pain (CPP). The study team is also interested in whether a web-based educational and self-management program for chronic pelvic pain changes how people think about chronic pelvic pain treatments. The program contains several different self-guided modules that include cognitive and behavioral structuring, self-administration of acupressure, engaging in physical activity, and a brief introduction to pelvic floor physical therapy techniques.

The study hypothesis is that patients with CPP will report that prior treatment experiences and most trusted source of medical information will be associated with baseline perceptions of various CPP treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic pelvic pain, defined as moderate to severe pelvic pain (based on protocol) for greater or equal to(≥) 6-month duration, and is non-cyclic, occurring for at least 14 days of each month.
* Must be scheduled for a new patient visit with the Chronic Pelvic Pain and Endometriosis Referral Clinic within the Department of Obstetrics and Gynecology at the University of Michigan for treatment of chronic pelvic pain.
* Access to internet via computer or smartphone
* English-language proficiency (current version of the website is in English)
* The study team will attempt to recruit a diverse group of patients, with attention to diversity in race, ethnicity, education level, rural vs urban locality, sexual orientation, and gender identification.

Exclusion Criteria:

* Severe physical impairment precluding participating in internet-based program (for example, complete blindness or deafness)
* Prior care within the Chronic Pelvic Pain and Endometriosis Referral Clinic within the Department of Obstetrics and Gynecology at the University of Michigan for treatment of chronic pelvic pain (seen previously but meets criteria for new patient visit because > 3 year interval since last clinic visit).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female sex assigned at birth, may include cis-gender, trans-gender, nonbinary
Enrollment: 30 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Explore factors that influence patient perceptions of treatment modalities for chronic pelvic pain | Baseline
  Explore prior treatment experiences, attitudes/perceptions of treatment modalities, sources of medical information. Baseline questionnaire and individual structured interview will be used.

SECONDARY OUTCOMES:
Change in self-reported interest in treatment modalities | Baseline, 3 weeks (post baseline)
  To evaluate whether brief exposure to a novel web-based educational and self-management program for chronic pelvic pain increases willingness to consider various treatment modalities one question will be asked.
  The question states are participants interested in trying six different treatment modalities and select from "yes, definitely interested", "would consider", "not sure, need to hear more about this option", or "not interested".
Change in credibility/expectancy questionnaire (CEQ) | Baseline, 3 weeks (post baseline)
  The CEQ is a self-report measure assessing the credibility and expectancy of treatment received. It consists of 6 items, 4 items with a 9-point Likert-type rating of 1 (not at all) to 5 (very much) with a scoring range of 3-27. The other 2 items are on a percentage scale from 0%-100% in increments of 10 with a scoring range of means 0-100%. Higher scores denote higher treatment credibility and expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Till, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT06540560/ICF_000.pdf